CLINICAL TRIAL: NCT02027870
Title: A Prospective Multicenter Single-Arm Observational Registry Study to Assess the Safety and Efficacy of EXCEL-II With Sirolimus Eluting Stent for the Treatment of Patients With de Novo Coronary Artery . (CREDIT-III Trial)
Brief Title: EXCEL-II DES to Treat the Patients With de Novo Coronary Artery Lesions. (CREDIT-III)
Acronym: CREDIT-III
Status: Completed | Type: Observational
Sponsor: JW Medical Systems Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CREDIT-III-131113
Record Dates: First submitted 2014-01-02; First posted 2014-01-06 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease
Keywords: DES; CAD; EXCEL-II; JWMS; PCI
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: None Retained — According to the CREATE (Multi - Center Registry of Excel Biodegradable Polymer Drug Eluting Stent) registration results show that ExcelTM drug-eluting stents implanted an average of 12 months, target lesion (TLF) the failure rate of 6.7%.Will this study expected target lesion group stent failure rate estimate of 6.7%, the target is 9.5%;Test hypothesis: bilateral 0.05% 0.05%, master degree, clinical follow-up requirements is more than 95%, this research need at least 829 patients, remove the CREDIT II randomized controlled study can provide the number of cases of test group 208 examples, this study still need to be included in the 621 patients.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- EXCEL-II DES: Using EXCEL-II biodegradable polymer sirolimus-eluting stent treating CAD
  Interventions: Device: EXCEL-II biodegradable polymer sirolimus-eluting stent

INTERVENTIONS:
Device: EXCEL-II biodegradable polymer sirolimus-eluting stent — EXCEL-II biodegradable polymer sirolimus-eluting stent implantation

SUMMARY:
The study aims to further assess the safety, efficacy and the performance of its delivery system of the new generation Sirolimus-eluting stent of JWMS up to five years.

DETAILED DESCRIPTION:
1. A prospective, a single set, multicenter clinical trial;
2. The primary in situ in patients with coronary heart disease;
3. The center of: 28 (the actual number of center shall prevail);The plan selected 621 patients;(where the total number of cases in 2.25 mm specification not less than 30 cases, 5 cases each specification of not less than 2.25 mm.)
4. Clinical follow-up time points: 1 months, 6 months, 12 months and 18 months of a year and 2 years to 5 years follow-up; This test by an independent coronary angiography core laboratories, data management and statistical center, clinical end points to judge committee and clinical monitoring of all relevant clinical and imaging data collecting, sorting, statistical analysis and judgement.All the selected patients within five years continuous follow-up tracking (phone or outpatient follow-up), to observe the happening of adverse events to the forward of the second generation of EXCEL drug-eluting stents (des) system security to make more accurate and credible evaluation.

ELIGIBILITY:
Inclusion criteria:

1.18yrs≤Age≤75yrs . 2..stability and unstable angina pectoris (AP), chronic myocardial infarction (OMI) or confirmed (myocardial ischemia; 3.De novo lesion at native coronary artery(Up to four target lesions). 4.Lesion length ≤60mm. 5.RVD 2.25mm～4.0mm. 6.DS%≥70% by visual estimation. 7.Coronary artery bypass surgery (coronary artery bypass grafting) patients. 8.Subjects are willing to follow the specified requirements follow-up.

9.To understand the purpose of testing, voluntary and signed informed consent, willing to accept the imaging and clinical follow-up of subjects.

Exclusion Criteria:

1. AMI within 7 days.
2. Left main lesion, transplant vasculopathy and stent restenosis lesion;
3. Severe calcified lesion unable to predilate.
4. The distortion of the stent was hampered by lesions.
5. NYHA≥Ⅲ or LVEF<35%.
6. Prior PCI within 1 year.
7. Pregnancy or lactation, and planning pregnancy or lactation.
8. Subjects have bleeding tendency or blood coagulation dysfunction or PCI contraindications, or anticoagulant therapy taboo or can't continue to take DAPT at least 1 year.
9. There are other diseases (such as cancer,malignant tumor ,congestive heart failure,organ transplantation or candidate) or abuse history (alcohol cocaine heroin, etc.), scheme compliance is poor, interference related data explanation or the limited life (< 1 year).
10. To aspirin heparin clopidogrel cobalt chromium alloy rapamycin PLA polymer contrast agent of one of allergy.
11. Serious liver and kidney function are not complete subject(ALT and AST were three times greater than the upper limit of normal).
12. Before enrolling to participate in other clinical trials and not reached the primary endpoint.
13. Non-compliant subject and could not finish the trial in accordance with the requirements of the subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the Patients With de Novo Coronary Artery Lesions
Sampling Method: Probability Sample
Enrollment: 625 (Actual)
Dates: Start 2014-01-08 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
The Target Lesion Failure(TLF) as the primary endpoint at 12-month | 12months
  Device-related cardiovascular composite endpoint, including cardiac death, target vessel MI and clinically driven TLR at 12 months post procedure

SECONDARY OUTCOMES:
Stent implantation success rate | 5 Years
TLF, cardiovascular composite endpoints, ARC defined stent thrombosis | 30 days, 6 months, and 2-5 years

CONTACTS AND LOCATIONS:
Overall Officials: yaling Han, MD, Principal Investigator — Shen yang Northern hospital
Locations (1):
- Shenyang Northern Hospital, Shenyang, Liaoning, China